CLINICAL TRIAL: NCT04039867
Title: Evaluation of Oxaliplatin and Gemcitabine in Patients With Metastatic Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was terminated due to halt in funding.
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, John P. Fruehauf, Professor of Clinical Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20043920; 20043920 (Other: University of California, Irvine); NCI-2011-01249 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2019-02-05; First posted 2019-07-31 (Actual); Results first posted 2020-01-02 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Carcinoma, Transitional Cell
Keywords: Carcinoma, Transitional Cell; Bladder Cancer; oxaliplatin; Gemcitabine
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Oxaliplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oxaliplatin with Gemcitabine (Experimental): Oxaliplatin will be given as an intravenous infusion over 60 minutes on Days 1 and 14 at a dose of 100 mg/m2 for each cycle. Gemcitabine (1000 mg/m2) will be given on days 1 and 14 as an intravenous infusion over 30 minutes immediately prior to Oxaliplatin.
  Interventions: Drug: Oxaliplatin with Gemcitabine

INTERVENTIONS:
Drug: Oxaliplatin with Gemcitabine — Oxaliplatin will be given as an intravenous infusion over 60 minutes on Days 1 and 14 at a dose of 100 mg/m2 for each cycle. Gemcitabine (1000 mg/m2) will be given on days 1 and 14 as an intravenous infusion over 30 minutes immediately prior to Oxaliplatin.
  Other Names: Gemzar; Eloxatin

SUMMARY:
This phase II trial evaluated the impact of Oxaliplatin and Gemcitabine in patients with recurrent or advanced transitional cell carcinoma of the bladder. The combination of Oxaliplatin and Gemcitabine is considered investigational and this study will help in determining if their activity and toxicity profiles are comparable or better than the standard regimens.

DETAILED DESCRIPTION:
The combination of Oxaliplatin and Gemcitabine has synergistic effects on a variety of human cancer cell lines in vitro. Clinically, it has demonstrated activity in other malignancies including lung, and pancreas. In the former study, poor prognosis advanced non-small cell lung cancer patients received Gemcitabine 1000mg/m2 and Oxaliplatin 65mg/m2 both on days 1 and 8. The overall response rate was 16%, with no reports of neutropenic fever. In the latter study, locally advanced and metastatic pancreatic cancer patients received Gemcitabine 1000mg/m2 on day 1 and Oxaliplatin 100mg/m2 on day 2 every 2 weeks. The overall response rate was 31%. The toxicity profile included grades 3 to 4 neutropenia and thrombocytopenia in 11%, 14% for nausea or vomiting, 6.2% for diarrhea, and 11% for peripheral neuropathy, with no toxic deaths

There has been one feasibility study evaluating the combination of Oxaliplatin and Gemcitabine in advanced transitional cell carcinoma (TCC) of the urothelium. Twenty patients with advanced urothelial carcinomas who were treated with Gemcitabine and Oxaliplatin at 1500mg/m2 and 85mg/m2 IV respectively, both on day 1 of a 14 day cycle. The median number of cycles was 5 and ranged from 1 to 7. A total of 90 cycles were delivered with 87 assessable for toxicity in 19 patients. No neutropenic fever occurred and G-CSF was not used although allowed as needed. Grades 3 to 4 neutropenia and thrombocytopenia were observed in 9 (10%) and 3 (3%) of the courses given respectively. Grades 1 to 2 neuropathy was noted to be common with only one patient suffering grade 3 neuropathy. Non-hematologic adverse effects were found to be mild. Response rates were not provided.

In summary, there is favorable evidence of antitumor activity in vitro and in clinical studies for a variety of cancers. Furthermore, the toxicity profile of this combination is also favorable. It is therefore logical to evaluate the effectiveness and tolerability of this combination in advanced urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically or cytologically confirmed diagnosis of transitional cell carcinoma of the bladder.
* Patients must have metastatic or locally recurrent transitional cell carcinoma of the bladder. Patients with locoregional disease must be considered incurable by means of locoregional therapy.
* All sites of disease must be assessed and designated as measurable or non- measurable disease as documented by CT, MRI, X-ray physical exam or nuclear exam. All measurable disease must be assessed within 28 days prior to registration. All non-measurable disease must be assessed within 42 days prior to registration.
* Patients must not have more than one prior chemotherapy regimen for recurrent/metastatic disease. Patients with initial locally advanced but nonmetastatic disease are allowed to have one prior chemotherapy regimen as part of the primary curative therapy. All chemotherapy must be completed 4 weeks prior to registration. Any number of prior biologic therapies (e.g. chimeric antibodies or kinase inhibitors) is permitted as part of the chemotherapy regimen.
* Patients may have received prior radiotherapy if there has been complete recovery from all radiation-induced toxicities. At least 4 weeks must have elapsed from the completion of radiation therapy to the time of registration. If lesions within the radiation port are to be used to assess response to therapy, those lesions must have demonstrated clear progression by the criteria outlined in Section 10.1.2V following completion of radiation therapy.
* Patients must not have a surgical procedure for bladder cancer within 4 weeks prior to registration. Patients must have completely recovered from all surgery prior to registration.
* Patients must have adequate bone marrow reserve as evidenced by ANC > 1,500 μl and platelets > 100,000/ μl obtained within 14 days prior to registration.
* Patients must have adequate hepatic function as evidenced by serum bilirubin <1.5x the institutional upper limit of normal. Serum transaminase (SGOT or SGPT) be must < 1.5 x the institutional upper limit of normal serum unless the liver is involved with tumor, in which case serum transaminase (SGOT or SGPT) must be < 5 x the institutional limit of normal. These tests must be obtained within 14 days prior to registration.
* Patients must have a creatinine < 2 x the institutional upper limit of normal obtained within 14 days prior to registration.
* All patients must be 18 years of age or older.
* Patients must have a Zubrod performance of 0-2.
* Patients must not have prior therapy with Oxaliplatin or Gemcitabine.

Exclusion Criteria

* Patients with severe psychiatric disorder are not eligible.
* Patients with known brain metastasis are not eligible. However, brain imaging studies are not required for eligibility if the patient has no neurological signs or symptoms. If brain imaging studies are performed, they must be negative for disease.
* No other prior malignancy is allowed except for adequately treated basal cell or squamous cell carcinoma, in situ cervical cancer, or adequately treated Stage I and II cancer from which the patient is in complete remission, or any other malignancy from which the patient has been disease-free for 5 years.
* Patients with any evidence of active or uncontrolled infection, recent myocardial infarction, unstable angina, or life-threatening arrhythmia are not eligible.
* Patients with any evidence of active or uncontrolled infection, recent myocardial infarction, unstable angina, or life-threatening arrhythmia are not eligible.
* Patients with severe psychiatric disorder are not eligible.
* Patients with known brain metastasis are not eligible. However, brain imaging studies are not required for eligibility if the patient has no neurological signs or symptoms. If brain imaging studies are performed, they must be negative for disease.
* No other prior malignancy is allowed except for adequately treated basal cell or squamous cell carcinoma, in situ cervical cancer, or adequately treated Stage I and II cancer from which the patient is in complete remission, or any other malignancy from which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-01-20 (Actual); Primary Completion 2011-10-06 (Actual); Study Completion 2011-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Fruehauf, MD, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxaliplatin With Gemcitabine
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eighteen patients were enrolled into the trial. There were 17 subjects that underwent treatment, with one dropping out before starting chemotherapy.
Arm/Group | Oxaliplatin With Gemcitabine
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 72 [58 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events to Evaluate Tolerability of Oxaliplatin With Gemcitabine
Description: To evaluate the tolerability of administering Oxaliplatin in combination with gemcitabine in patients with recurrent or advanced TCC bladder. Toxicity and adverse events are based on the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 3.0.
Time Frame: From date of registration until treatment completion, disease progression or other reasons for removal from protocol treatments, whichever came first, an average of 1 year.
Population: Please refer to the Adverse Event tables for specifics.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxaliplatin With Gemcitabine
Number analyzed (Participants) | 17
Participants | 17

2. Secondary Outcome: Overall Response Rate as Assessed by RECIST Criteria of Patients Who Received Gemcitabine and Oxaliplatin
Description: To assess the overall response rate to the combination of gemcitabine and Oxaliplatin in patients with recurrent or advanced TCC bladder. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI. Complete Response (CR) is defined as disappearance of all target lestions. Partial Response (PR) is defined as >=30% decrease in the sum of the longest diameter of target lesions. Overall response rate (ORR) is defined as confirmed complete response (CR) and partial response (PR). ORR = CR + PR
Time Frame: From date of registration until first date of disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 1 year.
Population: Only 14 were accessable for response. One subject never started treatment, two dropped out of the study and one died prior to first assessment.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin With Gemcitabine
Number analyzed (Participants) | 14
participants | 5

3. Secondary Outcome: Overall Survival of Patients Who Received Gemcitabine and Oxaliplatin
Description: To evaluate overall survival in patients with advanced TCC bladder treated with this combination of gemcitabine and Oxaliplatin.
Time Frame: From date of registration for 5 years or until death from any cause, whichever came first.
Population: All treated patients were included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oxaliplatin With Gemcitabine
Number analyzed (Participants) | 17
days | 314 [161.6 to 466.4]

ADVERSE EVENTS:
Time Frame: From date of registration until treatment completion, disease progression or other reasons for removal from protocol treatments, whichever came first, an average of 1 year.
Description: Toxicity was graded according to National Cancer Institute Common Terminology Criteria of Adverse Events, version 3.0. Safety was assessed through adverse event monitoring, physical examinations, vital signs and clinical laboratory tests before each dosing.
Arm/Group | Oxaliplatin With Gemcitabine
All-Cause Mortality (participants affected / at risk) | 10/17
Serious Adverse Events (participants affected / at risk) | 11/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin With Gemcitabine (N=17)
Anemia (Blood and lymphatic system disorders) | 2
Fatigue (General disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Sensory Neuropathy (Nervous system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin With Gemcitabine (N=17)
Anemia (Blood and lymphatic system disorders) | 6
Cold sensitivity (Nervous system disorders) | 4
Swelling (General disorders) | 6
Fatigue (General disorders) | 9
Sensory Neuropathy (Nervous system disorders) | 5
Nausea/vomiting (General disorders) | 10
Diarrhea (Gastrointestinal disorders) | 3
Anorexia (Psychiatric disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Injection Site Reaction (General disorders) | 4
Constipation (Gastrointestinal disorders) | 6
Chills (General disorders) | 3

LIMITATIONS AND CAVEATS:
The main limitation for our study was the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes